CLINICAL TRIAL: NCT04458948
Title: Open Label Non-comparative Trial of the Combination of Hydroxychloroquine and Azithromycin in the Treatment of Hospitalized Patients With Moderate or Severe COVID-19 Infection
Brief Title: Non-comparative Trial of the Combination of HCQ and AZI in the Treatment of ICU Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The World Health Organization (WHO) paused Hydrochloroquinone from its Solidarity Trial in order to conduct a safety data review by the Data Safety Monitoring Board of the WHO to evaluate HCQ in its clinical trials.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-156
Record Dates: First submitted 2020-06-09; First posted 2020-07-07 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydroxychloroquine and Azithromycin (Experimental): All subjects receive Hydroxychloroquine and Azithromycin.
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400 mg BID, on day 1 and then 200 mg BID day 2 through 7 IV or po for 5 days. If the condition of the patient does not allow for oral therapy, HCQ can be given via a feeding or NG tube. Azithromycin can be given intravenously.
Drug: Azithromycin — Azithromycin 500 mg, IV or po for 5 days

SUMMARY:
This research is designed as an open-label,non-comparative prospective trial.

DETAILED DESCRIPTION:
The objects of this research are as follows:

(1) To measure the duration of viral shedding in respiratory secretions of patients with moderate or severe COVID-19 infection treated with the combination of Hydroxychloroquine and azithromycin. (2) Evaluate the case fatality rate, the clinical response and length of stay in hospitalized patients with moderate and severe COVID-19 infection. (3) To report the safety of the drug combination in hospitalized patients with moderate and severe COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >18 years of age with lower respiratory infection with SARSCo2 documented by a positive RT-PCR in nasopharyngeal sample admitted to the University of New Mexico Hospital, with an oxygen saturation of less than 94%, on room air, or a respiratory rate >24 per minute, or HR>125 per minute of a PaO2/FIO2<150.
2. Patient with life expectancy >48 hours.
3. Pregnant women may be included if deemed necessary. There is insufficient information regarding the safety of hydroxychloroquine and azithromycin during pregnancy. Consequently, these medications are not recommended when pregnant or planning to become pregnant. However, investigators may prescribe hydroxychloroquine and azithromycin if deemed necessary.
4. Azithromycin is excreted in human milk, therefore participants should not breast-feed whilst taking Azithromycin, because it may cause side effects including diarrhoea and infection to a baby. It is recommended to discard the milk during treatment and up until 2 days after discontinuation of treatment. Additionally, hydroxychloroquine should not be taken whilst breast-feeding. However, investigators may prescribe hydroxychloroquine and azithromycin if deemed necessary. Page 6 of 23 Version Date: 04.16.2020
5. Adults unable to consent will be included with the consent of their Legally Authorized Representative (LAR). Assent will be pursued from cognitively impaired participants if they are able to provide assent. Note that this does not preclude the enrollment of cognitively impaired participants that cannot provide assent, but would allow those that can the opportunity to do so.

Exclusion Criteria:

1. Prisoners
2. Pre-/co-existing medical conditions, including any of the following:

   Known allergy to study drugs. Contraindication to treatment with study drugs, including retinopathy, and QTc prolongation defined by QTc>450 in males and >470 in females. Unless, it is the opinion of the treating physician(s) that the benefits to treat with medications outweigh the risks. Known chronic kidney disease, stage 4 or 5 or receiving dialysis. Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
3. Weight <40 kg.
4. Current use of: hydrocholoroquine or cardiac medicines of: flecainade, Tambocor; amiodarone Cordarone, Pacerone; digoxin or Digox, Digitek, Lanoxin; procainamide or Procan,Procanbid, propafenone, Rythmal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine and Azithromycin
Started | 28
Completed | 0
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: Our baseline population is from the state of New Mexico, Navajo nation and other surrounding Pueblo nations. We enrolled 28 patients, about equal males and females, ages from 32 to 85.
Groups:
- ICU Patients in Our Quarterary Care: 28 individuals admitted with severe COVID-19 pneumonia.
Arm/Group | ICU Patients in Our Quarterary Care
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 19
Age, Continuous [Mean (Full Range); unit: years] | 70 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had Viral Shedding as Determined by RT-PCR.
Description: To measure the duration of viral shedding in respiratory secretions of patients with moderate to severe COVID-19 infection treated with the combination of Hydroxychloroquine and azithromycin.
Time Frame: 14 to 28 days.
Population: 28 patients all had COVID -19 pneumonia.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 28
Participants | 6

ADVERSE EVENTS:
Time Frame: Days 1-5 of admission.
Description: Adverse events were not related to drug intervention.
Arm/Group | Hydroxychloroquine and Azithromycin
All-Cause Mortality (participants affected / at risk) | 28/28
Serious Adverse Events (participants affected / at risk) | 9/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine and Azithromycin (N=28)
Clotting to vital organs (lungs, heart, kidney and brain) (Respiratory, thoracic and mediastinal disorders) | 9 (9) — All patients passed at one month. 9 passed during day 1 to 5 of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04458948/Prot_004.pdf
  • Informed Consent Form (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04458948/ICF_005.pdf